CLINICAL TRIAL: NCT07006194
Title: Nicotinamide Levels in Serum, Aqueous Humor, and Tear Film in Glaucoma and Correlations With Mitochondrial Damage-Associated Molecular Patterns (mtDAMPs) and Senescence-Associated Secretory Phenotype (SASP)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi 'G. d'Annunzio' Chieti e Pescara (Other)
Collaborators: OFFHEALTH S.p.A. (Industry); Università degli Studi di Sassari (Other); University of Pisa (Other)
Responsible Party: Principal Investigator, Luca Agnifili, Associate Professor, Università degli Studi 'G. d'Annunzio' Chieti e Pescara
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: NAD-mtDAMPs-SASP
Record Dates: First submitted 2025-02-24; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Glaucoma
Keywords: glaucoma; Nicotinamide; mtDAMPs; SASP; aqueous humor; tear film; senescence
MeSH Terms: conditions — Glaucoma | interventions — Niacinamide

STUDY DESIGN:
Intervention Model Description: Tricentric case-control cross-sectional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- OAG not pharmacologically controlled, receiving MTM and scheduled for filtering glaucoma surgery (No Intervention): Patients with open-angle glaucoma (OAG) not pharmacologically controlled, receiving maximal tolerated medical therapy and scheduled for filtering glaucoma surgery (stand-alone or combined). To this arm will be administered ophthalmological evaluation, functional stage determination, OCT imaging, sampling and analysis of biological fluids (Plasma and Peripheral Blood Mononuclear Cells (PBMCs) Isolation, Tear Film, Aqueous Humor; NAD Quantification in all biological fluids, mtDAMPS and SASP quantification in PBMCs)
- Pharmacologically controlled OAG scheduled for cataract surgery (No Intervention): Patients with pharmacologically controlled OAG scheduled for cataract surgery. To this arm will be administered ophthalmological evaluation, functional stage determination, OCT imaging, sampling and analysis of biological fluids (Plasma and Peripheral Blood Mononuclear Cells (PBMCs) Isolation, Tear Film, Aqueous Humor; NAD Quantification in all biological fluids, mtDAMPS and SASP quantification in PBMCs)
- Healthy individuals scheduled for cataract surgery (No Intervention): Healthy individuals scheduled for cataract surgery. To this arm will be administered ophthalmological evaluation, functional stage determination, OCT imaging, sampling and analysis of biological fluids (Plasma and Peripheral Blood Mononuclear Cells (PBMCs) Isolation, Tear Film, Aqueous Humor; NAD Quantification in all biological fluids, mtDAMPS and SASP quantification in PBMCs)
- Pharmacologically controlled OAG patients scheduled for cataract surgery and treated with iNAD (Experimental): Pharmacologically controlled OAG patients scheduled for cataract surgery and treated with iNAD. To this arm will be administered iNAD during the month preceding surgery and ophthalmological evaluation, functional stage determination, OCT imaging, sampling and analysis of biological fluids (Plasma and Peripheral Blood Mononuclear Cells (PBMCs) Isolation, Tear Film, Aqueous Humor; NAD Quantification in all biological fluids, mtDAMPS and SASP quantification in PBMCs)
  Interventions: Dietary Supplement: Nicotinamide Tablet

INTERVENTIONS:
Dietary Supplement: Nicotinamide Tablet — One nicotinamide tablet per day during the month preceding surgery
  Arms: Pharmacologically controlled OAG patients scheduled for cataract surgery and treated with iNAD

SUMMARY:
Background Glaucoma is a multifactorial, chronic, and progressive eye disease characterized by the irreversible loss of retinal ganglion cells (RGCs). It is the second leading cause of blindness globally, with approximately 76 million patients affected in 2020, a number expected to rise to 120 million in the coming decades, especially in Africa and Asia. Elevated intraocular pressure (IOP) is a significant risk factor for glaucoma, and its reduction remains the only scientifically proven approach to slowing visual function decline. However, many glaucoma patients continue to experience visual loss even with IOP values within the normal range, due to the disease's multifactorial nature. Besides IOP reduction, there is a need for direct neuroprotection to address other factors causing RGC damage.

Mitochondrial dysfunction has emerged as a critical early factor in RGC damage, making glaucoma, at least in part, resemble a mitochondrial disease. Mitochondria play a key role in cellular functions such as energy production, redox metabolism, and maintaining mitochondrial function. In glaucomatous conditions, mitochondrial damage leads to the release of mitochondrial damage-associated molecular patterns (mtDAMPs), triggering chronic inflammation and tissue damage. This inflammation is exacerbated by the Senescence-Associated Secretory Phenotype (SASP), a process where senescent cells secrete bioactive molecules that contribute to cellular dysfunction and glaucoma progression.

Among potential neuroprotective approaches, nicotinamide (NAM) and its precursor nicotinamide riboside (NR) are gaining attention. These compounds support mitochondrial function and NAD production, which is essential for cellular vitality. Research indicates that reductions in NAM levels correlate with glaucoma progression. For instance, studies have shown that NAD precursors may prevent or delay RGC degeneration, suggesting a promising adjunctive treatment for glaucoma patients.

Study Objectives The study aims to measure NAM levels in ocular and non-ocular biological fluids (serum, aqueous humor, and tear fluid) of patients at different stages of glaucoma. The study will correlate NAM concentrations with disease severity and mitochondrial function markers. Furthermore, NAD levels in peripheral blood mononuclear cells (PBMCs) will be assessed to investigate potential biomarkers for glaucoma progression. A secondary objective is to evaluate the impact of dietary supplementation with nicotinamide and nicotinamide riboside (iNAD®) on NAD levels in pharmacologically controlled glaucoma patients.

Methods This cross-sectional, case-control, multi-center study involves three universities: University of G. d'Annunzio Chieti-Pescara, University of Pisa, and University of Sassari. Biological fluid analyses will be conducted at the Animal Biology Laboratory affiliated with the University of G. d'Annunzio Chieti-Pescara.

Patients will be categorized into four groups:

1. Uncontrolled glaucoma patients scheduled for glaucoma surgery.
2. Controlled glaucoma patients scheduled for cataract surgery.
3. Healthy controls undergoing cataract surgery.
4. Pharmacologically controlled glaucoma patients supplemented with iNAD®. Biological fluids (plasma, PBMCs, tear fluid, and aqueous humor) will be collected for analysis, including measures of NAD, mtDAMPs, and SASP components. These measures aim to provide insights into the molecular mechanisms underlying glaucoma and potential biomarkers for disease progression.

Statistical Analysis Sample size estimation was calculated using G*Power for a priori one-way ANOVA analysis. Assuming a mean NAM concentration of 0.14 μM (SD=0.12) for glaucoma patients and 0.19 μM (SD=0.13) for controls, with a power of 80% and alpha of 0.05, a minimum of 246 patients (82 per group) are required.

DETAILED DESCRIPTION:
Background Glaucoma is a multifactorial, chronic, and progressive disease characterized by the irreversible loss of retinal ganglion cells (RGCs). It represents the second leading cause of blindness globally, but it is the leading cause of irreversible blindness, with 76 million patients affected worldwide in 2020. Unfortunately, it is estimated that the incidence of the disease will increase significantly in the next two decades, with approximately 120 million patients affected globally, particularly in Africa and Asia. Elevated intraocular pressure (IOP) is one of the most important risk factors for the development and progression of the disease, and its reduction is the only scientifically proven approach to controlling the decline in visual function. However, despite the reduction in IOP slowing the worsening of visual fields, many glaucoma patients continue to experience progressive loss of visual function despite IOP values within the statistical normal range. This is because glaucoma is a multifactorial disease, and simply reducing IOP does not guarantee the control of other risk factors damaging RGCs.

Among the mechanisms involved in the damage and death of RGCs in glaucoma, mitochondrial dysfunction appears to be one of the most important and earliest, leading the scientific literature to consider glaucoma, at least in part, as a particular form of mitochondrial disease. The need for direct neuroprotection, in addition to indirect neuroprotection (IOP reduction), represents a significant unmet need in the management of glaucoma patients. At present, despite numerous preclinical and some clinical evidence supporting the efficacy of certain molecules (such as citicoline) in protecting RGCs, there is no scientifically supported neuroprotective therapy in humans.

Two forms of vitamin B3, nicotinamide (NAM) and nicotinamide riboside (NR), are emerging as potential adjunctive therapies for the protection and enhancement of RGCs. These compounds are precursors to nicotinamide adenine dinucleotide (NAD). NAD is essential for the proper functioning of cells and is involved in various metabolic activities, including energy production, acting as a key cofactor in redox metabolism, including glycolysis, the citric acid cycle, oxidative phosphorylation, protection against reactive oxygen species, contributing to various enzymatic activities, and maintaining mitochondrial function.

Mitochondria, traditionally recognized for their role in bioenergy production and metabolite generation, are gaining increasing recognition for their various functions, including cellular signaling, cell death, regulation of reactive oxygen species (ROS), and inflammation. Given the high susceptibility of RGCs to mitochondrial damage, mitochondrial dysfunction becomes intricately linked to a series of cellular processes (aging, excitotoxicity, oxidative stress, mitophagy deficiency, prolonged inflammatory responses) associated with the pathogenesis of glaucoma. In glaucomatous conditions, the removal of defective mitochondria becomes crucial for maintaining mitochondrial quality control, thereby protecting cellular integrity. Consequently, mitochondrial dynamics, biogenesis, and mitophagy play crucial roles in ensuring effective mitochondrial quality control. Mitochondrial damage in neurons, particularly in RGCs, leads to the release of "Mitochondrial damage-associated molecular patterns" (mtDAMPs). These molecules act as triggers for chronic inflammation through pattern recognition receptors (PRRs) on glial cells and complementary activations in glaucoma. Numerous mtDAMPs, including mtDNA, ATP, cardiolipin, mitochondrial transcription factor A (TFAM), N-formyl peptides (NFPs), and cytochrome c, have been implicated in inducing an inflammatory process. The immunogenic nature of mtDNA, similar to bacterial DNA, activates interferon (IFN)-dependent genes, TLR9, the NLRP3 inflammasome, and the cGAS-STING signaling pathway. Defects in mitochondrial synthesis and maintenance, as well as alterations in mitophagy (autophagy of mitochondria), can contribute to dysfunctional accumulation, compromising energy (ATP) production and cellular metabolism regulation. These alterations can negatively impact cellular vitality and functionality, promoting cellular senescence. Emerging evidence suggests a link between glaucomatous conditions and cellular senescence. RGC senescence may contribute to the pathogenesis of glaucoma. The accumulation of senescent cells in the eye could lead to disrupted tissue homeostasis and compromised cellular function, potentially worsening glaucoma progression. Senescent cells can secrete a variety of bioactive molecules, a phenomenon known as Senescence-Associated Secretory Phenotype (SASP). SASP components released into bodily fluids include cytokines, chemokines, growth factors, and extracellular matrix remodeling enzymes. These factors can act in a paracrine manner, influencing nearby cells and contributing to chronic inflammation and tissue malfunction. In glaucoma, the presence of SASP components in biological fluids may indicate a dynamic interaction between senescent cells and the surrounding microenvironment. Understanding the presence and impact of senescence and SASP in biological fluids is crucial for unraveling the complex molecular mechanisms underlying glaucoma progression.

Emerging evidence has demonstrated that axonal degeneration in glaucomatous cells is associated with a decline in NAD, and the supplementation of NAD or NAD precursors (NAM or NR) may be effective in preventing or delaying RGC death in vitro and in vivo. In an experimental study, Williams and colleagues showed that oral administration of NAM was able to increase NAD levels in the retina and protect RGCs from degeneration in a murine glaucoma model. Interestingly, 93% of the experimental animals supplemented orally with a high dose of NAM (2000 mg/kg/day) did not develop RGC loss despite high IOP. Given its beneficial effects and evidence of reduced NAD bioavailability with aging, numerous research directions are exploring ways to restore cellular NAD pools in humans by administering its precursors.

Study Objectives Initial evidence has indicated a reduction in NAM concentrations by over 30% in the serum of glaucoma patients. However, no studies have been conducted to assess NAM levels in ocular biological fluids of patients with glaucoma at various stages of the disease.

The tear film, potentially rich in intraocular-derived molecules (due to trans-scleral flows of aqueous humor), and the aqueous humor itself, which directly bathes the sensitive sites of the disease (e.g., trabecular meshwork), are likely to express more significant and glaucoma-specific variations in NAM concentrations compared to those detectable in plasma or other distant fluids.

Studying ocular and non-ocular biological fluids can provide valuable insights into the molecular landscape associated with glaucoma. Analyzing these fluids for specific SASP markers, inflammatory cytokines, and molecules associated with mitochondrial dysfunction could reveal potential diagnostic and prognostic indicators for glaucoma progression.

Recent research has shown that in peripheral blood mononuclear cells (PBMC) from POAG patients, there is a reduction in mitochondrial respiration and NAD levels, and the degree of mitochondrial impairment correlates with the likelihood of glaucoma progression. In the same study, NAD levels in PBMC are proposed as a clinical diagnostic biomarker for glaucoma progression. Given various clinical studies investigating the effects of dietary supplementation with nicotinamide metabolic precursors on glaucoma progression, it is essential to demonstrate the impact of such treatments on NAD levels in PBMC among POAG patients.

Monitoring variations in senescence-associated molecules, alongside mitochondrial dysfunction linked to nicotinamide, could offer a non-invasive method to evaluate the severity and progression of the disease, enabling early interventions and personalized treatment strategies.

Main Outcomes:

1. Measure NAM levels in serum, aqueous humor, and tear fluid in open-angle glaucoma (POAG): i) in patients with decompensated glaucoma candidates for glaucoma surgery; ii) in patients with pharmacologically controlled glaucoma candidates for cataract surgery; iii) and in healthy controls candidates for cataract surgery.
2. Correlate NAM concentrations in the three fluids with disease stage, assessed through MD and VFI (Hodapp classification for staging) and RoP (if available).
3. Correlate NAM levels with mitochondrial function indicators (mtDAMPs).
4. Measure NAD content in PBMCs from the aforementioned patient cohorts.
5. Measure NAD content in PBMCs from pharmacologically controlled POAG patients at baseline and after one month of dietary supplementation with a product containing nicotinamide and nicotinamide riboside (iNAD®).

Secondary Outcomes:

1. Correlate NAM concentrations with pre-surgery IOP levels and baseline levels.
2. Correlate NAD concentrations in aqueous humor with NAM levels in tear fluid and plasma.
3. Assess if there is a different NAD concentration in primary and secondary (PEX/PG) open-angle glaucoma.
4. Correlate NAD levels with SASP components. Methods Study Design This is a cross-sectional, case-control, multi-center study involving the University of G. d'Annunzio Chieti-Pescara (Prof. Luca Agnifili), the University of Pisa (Prof. Michele Figus), and the University of Sassari (Prof. Matteo Sacchi). The ophthalmology departments of the three universities will be responsible for patient enrollment, diagnostic and surgical procedures, and biological fluid sampling.

Biological fluid analyses will be conducted at the Animal Biology Laboratory (Body C, Level 1, Pharmacy Building) affiliated with the Biomorphology section of the Department of Medicine and Aging Sciences at the University of G. d'Annunzio Chieti-Pescara (Head: Prof. Antonia Patruno).

Patients

The study will recruit:

* 90 patients with open-angle glaucoma (OAG) not pharmacologically controlled, receiving maximal tolerated medical therapy and scheduled for filtering glaucoma surgery (stand-alone or combined) (Group 1).
* 90 patients with pharmacologically controlled OAG scheduled for cataract surgery (Group 2).
* 90 healthy individuals scheduled for cataract surgery (Group 3).
* 90 pharmacologically controlled OAG patients scheduled for cataract surgery and treated with iNAD (Group 4).

Before enrollment, each patient will sign an informed consent form outlining the nature and potential consequences of the study.

Procedures

1. Ophthalmological Evaluation A complete ophthalmological evaluation will be conducted at enrollment, including best-corrected visual acuity, optical pachymetry using AS-OCT (CIRRUS HD-OCT 5000, ZEISS, Dublin, CA), Goldmann tonometry (three measurements between 8-10 am and 4 pm), gonioscopy, anterior and posterior segment analysis (in mydriasis) using slit lamp examination.
2. Functional Stage Determination The glaucoma stage will be determined by measuring the mean defect (MD, dB) using standard automated perimetry (HFA; Carl Zeiss Meditec, Dublin, CA, USA) with the 24-2 SITA-Fast strategy. Defects will be classified according to Hodapp-Parrish-Anderson criteria: mild (MD > -6 dB), moderate (MD between -6 dB and -12 dB), advanced (MD < -12 dB), and severe (MD < -20 dB with central fixation loss). For patients with a sufficient number of visual fields performed on the same platform, a rate of progression will be calculated using trend analysis (GPA; HFA; Carl Zeiss Meditec, Dublin, CA, USA).
3. OCT Imaging OCT measurements for average and sectoral RNFL and GCC thickness will be performed using the Cirrus platform.

Sampling of Biological Fluids Biological fluids will be collected simultaneously on the same day as the surgical procedure in the morning while fasting.

1. Plasma and Peripheral Blood Mononuclear Cells (PBMCs) Isolation Blood samples will be collected in heparin tubes. Immediately after collection, tubes will be transported on ice to the Animal Biology Laboratory (Body C, Level 1, Pharmacy Building) at the University of G. d'Annunzio Chieti-Pescara (Head: Prof. Antonia Patruno), where PBMC isolation and plasma recovery will be performed.

   For participants at the two off-site ophthalmology units, blood samples will be collected in heparin tubes and treated with an appropriate volume of TransFix® (200 µL TransFix® per 1000 µL of blood, 1:5 ratio). Blood treated with TransFix® may be stored for up to 14 days at 2-8°C, suitable for transfer to the Animal Biology Laboratory at the University of G. d'Annunzio Chieti-Pescara.

   PBMCs will be separated from other components by centrifugation for 30 minutes at 1500 rpm using a density gradient with Ficoll-Paque (density: 1.007 g/mL). Red blood cells, granulocytes, and dead cells will pass through the Ficoll layer, while lymphocytes and monocytes will accumulate at the plasma-Ficoll interface forming a cell ring. The plasma will be collected in a 1:1 ratio with PBS and gently mixed with Ficoll in a 1:1 ratio. Following centrifugation at 1500 rpm for 30 minutes at 22°C, plasma will be collected and stored at -80°C.

   The PBMC cell ring will be washed twice with PBS to remove the supernatant and resuspended in QIAzol (lysis reagent, QIAGEN Sciences, MD, USA) for RNA isolation, then frozen at -80°C.
2. Tear Film Tear samples will be obtained using a Schirmer strip inserted into the inferior conjunctival sac for 5 minutes with eyes closed. Each Schirmer strip will be placed in an Eppendorf tube and transported on ice to the Animal Biology Laboratory (Body C, Level 1, Pharmacy Building) at the University of G. d'Annunzio Chieti-Pescara (Head: Prof. Antonia Patruno), where the tear film recovery protocol will be performed.

   For off-site ophthalmology units, tear samples will be stored at -20°C and transferred on dry ice to the Animal Biology Laboratory.

   Tear film recovery: Each Schirmer strip soaked with tears will be placed in 70 µL of T-PER (Tissue Protein Extraction Reagent, Pierce) at room temperature for 2 hours. The Schirmer strip will then be collected and centrifuged at 4°C at 13,000 g for 2 minutes. The tear solution (80±5µL, 1.5±0.5µg µL-1) will be divided into aliquots and stored at -80°C.
3. Aqueous Humor Aqueous humor (0.5 - 1 ml) will be collected immediately and carefully at the beginning of surgery, prior to any surgical steps, via anterior chamber paracentesis using a 27-gauge needle connected to a tuberculin syringe under a surgical microscope. During this procedure, intraocular tissues such as the iris and lens will be carefully avoided. The aqueous humor will be immediately transferred to the Animal Biology Laboratory (Body C, Level 1, Pharmacy Building) at the University of G. d'Annunzio Chieti-Pescara (Head: Prof. Antonia Patruno) and stored at -80°C until all tests are performed. All samples will be protected from light.

   For off-site units, samples will be stored at -20°C and transferred on dry ice to the Animal Biology Laboratory.
4. NAD Quantification Total NAD (NAD and NADH) will be quantified using a spectrophotometric assay with a reference wavelength of 450 nm.
5. mtDAMPS Analysis

   1. Extraction of nucleic acids: Isolation of mtDNA from biological samples.
   2. ATP levels will be measured using luminometric techniques.
   3. Cardiolipin levels will be assessed using chromatography techniques.
   4. TFAM levels will be evaluated through immunoprecipitation techniques.
   5. Detection of formylated peptides (NFPs) using mass spectrometry.
   6. Cytochrome c levels will be measured via immuno-enzymatic techniques.
6. SASP Measurement Quantitative analysis of specific SASP components (e.g., IL-6, IL-8, MMPs, PAI-1) will be performed using immuno-enzymatic techniques (ELISA). Results validation will be done via Western blot to identify specific SASP proteins.

Statistical Analysis.

ELIGIBILITY:
Group 1 Inclusion Criteria

* Age > 18 years
* Diagnosis of open-angle glaucoma (primary open-angle glaucoma)
* Uncontrolled IOP (> 21 mmHg as the mean of three measurements between 8-10 am and 16),
* Maximal medical therapy
* Perimetric-OCT and ophthalmic optic neuropathy criteria
* Indication for standalone or combined glaucoma surgery (any surgery allowing aqueous humor sampling: MIGS, MIBS, TRABE, DS, canal surgery, drainage tube implants, revision of surgical implant)

Group 2 and 4 Inclusion Criteria

* Age > 18 years
* Diagnosis of open-angle glaucoma
* Controlled IOP (≤ 21 mmHg as the mean of three measurements between 8-10 am and 16) under medical therapy (excluding oral acetazolamide)
* Perimetric-OCT and ophthalmic optic neuropathy criteria.

Group 3 Inclusion Criteria:

* Age >18 years
* IOP ≤ 21 mmHg
* Absence of perimetric-OCT and ophthalmic optic neuropathy criteria for glaucoma.

Exclusion Criteria for all groups

* Conditions and systemic therapies influencing NAM levels in biological fluids
* Concomitant ocular pathologies beyond glaucoma or cataracts
* Ocular therapies beyond hypotensive eye drops
* Prior ocular surgeries
* Secondary glaucomas (uveitic, silicone oil, traumatic, neovascular)
* End-stage glaucoma or severe glaucoma (<-20 dB)
* Pregnancy and breastfeeding.
* (only for Group 3) family history of glaucoma and transient IOP spikes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Nicotinamide levels measurement in biologic fluids | Day 1
  Measure nicotinamide levels in serum, aqueous humor, and tear fluid in open-angle glaucoma (POAG): i) in patients with decompensated glaucoma candidates for glaucoma surgery; ii) in patients with pharmacologically controlled glaucoma candidates for cataract surgery; iii) and in healthy controls candidates for cataract surgery.
Nicotinamide levels clinical correlation | Day 1
  Correlate NAM concentrations in the three fluids with disease stage, assessed through MD and VFI (Hodapp classification for staging) and RoP (if available).
Nicotinamide levels - mtDAMPs correlation | Day 1
  Correlate NAM levels with mitochondrial function indicators (mtDAMPs).
Nicotinamide levels measurement in PBMCs | Day 1
  Measure NAD content in PBMCs
Nicotinamide levels measurement after dietary supplementation | At enrollment and at the end of treatment at 4 weeks
  Measure NAD content in PBMCs from pharmacologically controlled POAG patients at baseline and after 4 weeks of dietary supplementation with a product containing nicotinamide riboside

SECONDARY OUTCOMES:
Nicotinamide levels - IOP correlation | Day 1
  Correlate NAM concentrations with pre-surgery IOP levels and baseline levels.
Nicotinamide levels in different biological fluids correlation | Day 1
  Correlate NAD concentrations in aqueous humor with NAM levels in tear fluid and plasma
Nicotinamide levels in different OAG types | Day 1
  Assess if there is a different NAD concentration in primary and secondary (PEX/PG) open-angle glaucoma
Nicotinamide levels - SASP correlation | Day 1
  Correlate NAD levels with SASP components

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Clinica Oftalmologica - Ospedale Clinicizzato SS Annunziata di Chieti, Chieti Scalo, Chieti
  - U.O. Oculistica Universitaria, Pisa, Pisa
  - Clinica Oculistica AOU Sassari, Sassari, Sassari